CLINICAL TRIAL: NCT04827524
Title: Investigation of Anthropometric Properties of Babies With Craniosynostosis
Status: Completed | Type: Observational
Sponsor: Yuksek Ihtisas University (Other)
Responsible Party: Principal Investigator, Melek Volkan Yazici, Principal Investigator, Yuksek Ihtisas University
Other Study IDs: Craniosynostosis
Record Dates: First submitted 2021-03-31; First posted 2021-04-01 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Craniosynostoses
MeSH Terms: conditions — Craniosynostoses

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Anthropometric measurement — The demographic information and birth histories of the subjects included in the study will be taken first. Anthropometric measurements of all subjects will be measured with the Star Scanner device. The Star Scanner 3 dimensional data collection system is a scanning system that enables the anthropometric head measurements of the baby to be taken in just 2 seconds. The advantages of this device is that it does not emit any harmful beams during evaluation, it does not have any harmful effects on health, and that it is an application that will not disturb babies.

SUMMARY:
Craniosynostosis is a malformation affecting the head and face, in which one or more sutures in the skull are fused prematurely. Premature union of one or more sutures causes changes in the shape of the skull base and dome, resulting in asymmetrical or restricted head and facial enlargement. It has been reported that in craniosynostosis, the bone enlargement is perpendicular to the fused sutures with the counterbalancing expansion. Craniosynostosis usually involves the union of a single cranial suture, but in some cases it has been observed that it may involve more than one suture in the baby's skull. An asymmetrical appearance is observed on the faces of babies, especially an unusual appearance in the form of eyes and skulls. It may present with neurological defects such as hydrocephalus, mental retardation, vision and hearing loss, as well as cosmetic deformities in the skull and facial bones. The general prevalence of craniosynostosis is around 1/2500 births. Generally, in single suture synostoses, there is no clear neurological finding except deformity. In multisuture synostoses there are a wide spectrum of findings such as increased intracranial pressure, hydrocephalus, syringomyelia, Chiari malformation, venous anomalies, ophthalmologic problems, growth retardation and epilepsy. Early diagnosis and treatment provides enough room for the baby's brain to grow and develop. It is thought that by measuring the anthropometric properties of these babies, the course of their development will be examined.

DETAILED DESCRIPTION:
Babies diagnosed with craniosynostosis at birth will be included in this study. The patients will be diagnosed using a combination of physical examination, skull radiographs and 3 dimensional computerized tomography scans.A voluntary consent form will be signed by the parents of all subjects indicating that they are willing to participate in the study. Anthropometric measurements of all subjects will be measured with the Star Scanner device.

ELIGIBILITY:
Inclusion Criteria:

* Being under 2 years old
* Being diagnosed with non-syndromic craniosynostosis
* Agreeing to participate in the study

Exclusion Criteria:

* Having a craniomaxillofacial fracture
* Having a history of surgery
* Having a congenital anomaly that affects growth or development

Ages: 1 Month to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: -Babies diagnosed with craniosynostosis at birth will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
3 dimensional anthropometric analysis of the cranium | Change from baseline anthropometric measure at 3 months.
  The 3 dimensional anthropometric analysis of the subjects cranium wil be measured using the Star Scanner device.

CONTACTS AND LOCATIONS:
Overall Officials: Melek Volkan-Yazici, PhD, Principal Investigator — Yuksek Ihtisas University
Locations (1):
- Yuksek Ihtisas University, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to ethical reasons.